CLINICAL TRIAL: NCT06096428
Title: The Assessment of Intravascular Peri-procedural Hemolysis During Catheter Ablation for Atrial Fibrillation Using Radiofrequency and Pulsed-field Energy
Brief Title: Hemolysis During Pulsed-field and Radiofrequency Ablation
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Charles University, Czech Republic (Other)
Responsible Party: Sponsor
Other Study IDs: PFA HEMOLYSIS
Record Dates: First submitted 2023-09-20; First posted 2023-10-23 (Actual); Last update posted 2023-11-15 (Actual); Status verified 2023-09

CONDITIONS: Atrial Fibrillation; Hemolysis; Pulsed-field Ablation
MeSH Terms: conditions — Atrial Fibrillation; Hemolysis | interventions — Radiofrequency Ablation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood drawing for hemolysis assessment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pulsed-field group: Patients will undergo catheter ablation for atrial fibrillation using pulsed-field energy
  Interventions: Device: Pulsed-field ablation
- Radiofrequency group: Patients will undergo catheter ablation using radiofrequency energx
  Interventions: Device: Radiofrequency ablation

INTERVENTIONS:
Device: Pulsed-field ablation — Pulsed-field ablation will be done using pentaspline catheter (Farawave, Boston Scientific) and pulsed-field energy generator. The goal will be achieve of electrical isolation of pulmonary veins.
  Groups: Pulsed-field group
Device: Radiofrequency ablation — Pulmonary vein isolation will be done using radiofrequency catheter (Qdot, Biosense-Webster) and generator of radiofrequency energy (nGEN, Biosense-Webster).
  Groups: Radiofrequency group

SUMMARY:
Hemolysis during and after catheter ablation will be compared between catheter ablation performed using radiofrequency and pulsed-field energy. Consecutive patients indicated for catheter ablation for AF will be enrolled, catheter ablation will be done using standard catheters (Qdot, Biosense Webster for RF, and Farapulse, Boston-Scientific for PF). Blood samples will be drawn at the beginning of ablation (T1), at the end of ablation (T2), and one day after the procedure (T3). Hemolysis will be analyzed using flow cytometry, ELISA and standard biochemistry and compared between RF and PF patients, Primary hypothesis is that hemolysis level will be higher after PF ablation compared to RF ablation.

DETAILED DESCRIPTION:
Catheter ablation presents the most effective treatment for atrial fibrillation (AF). It consists of the electrical isolation of the pulmonary veins. Several kinds of ablation energies can be used for the ablation. So far, the most often kind of energy was radiofrequency (RF) energy that leads to thermal destruction of the cardiac tissue. Newly, pulsed-field (PF) energy was developed for catheter ablation of AF. The use of PF energy consists in ultra-short, high-power application of electrical impulses that lead to fast, non-thermal cardiac tissue destruction.

Despite significant advantages, such as tissue selectivity, short procedure duration, and high durability of ablated lesions, the use of PF energy could also have other adverse effects. Recently, renal failure due to accelerated peri-procedural hemolysis in patients with pre-existed renal disease was described after PF ablation for AF.

The aim of the project is to assess and compare the level of hemolysis during catheter ablation for AF using PF and RF energy. Sixty consecutive patients indicated for catheter ablation for AF according to the standard recommendation (symptomatic paroxysmal or non-paroxysmal AF) will be enrolled. Consecutive patients as they are scheduler for procedure will be enrolled without randomization. In 40 patients (20 paroxysmal and 20 non-paroxysmal), the ablation will be done using PF energy, and in 20 patients using RF energy.

In all patients, intracardiac echocardiography (Accunav, Siemens, Germany) and fluoroscopy will be used for navigation. The procedures will be done as it is currently routinely done in the EP lab. In RF patients, 4 vascular access will be used (one for 10-pole catheter placed into the coronary sinus, one for intracardiac echocardiography probe, and 2 for transseptal sheaths). Two transseptal punctures will be done under the guidance of intracardiac echocardiography using SL1 sheaths (Abbott, USA). One transseptal access will be used for diagnostic circular mapping catheter (Lasso, Biosense-Webster, USA), the other for the ablation catheter. The RF ablation will be performed using SmartTouch or QDot ablation catheters (both Biosense-Webster, USA); however, ablation will be driven by the ablation index even if QDot catheter is used. The RF ablation will be performed using ablation index (400-450 on anterior-superior aspects and 350-400 on posterior aspects of PVs), the QDot Plus (high-power short-duration) regimen won´t be used. The goal will be to achieve the entrance and exit block of all 4 PVs. In non-paroxysmal patients, additional ablations could be done at the discretion of the treating physician (fractionated singnals, lines).

In the PF patients, two vascular access will be obtained. The first will be used for intracardiac echocardiography, the second for the transseptal sheath. Transseptal puncture will be done also using SL1 sheath (Abbott, USA), and using over-the-wire technique, this sheath will be exchanged by the 16-F Faradrive sheath (BSCI, USA). The ablation then will be done using pentaspline ablation catheter (Farawave, Boston Scientific). Four application of pulsed-field energy in basket configuration, and 4 application in flower configuration will be applied to each pulmonary vein. Additional pulsed-field energy application could be added if the signal in PV are present. In non-paroxysmal patients, additional pulsed-field energy application could be applied on the discretion of the operator on the posterior wall, or mitral isthmus.

Blood samples will be taken at the beginning of the procedure from the femoral vein (T1), at the end of the procedure after ablation lesions completion (T2), and one day after the procedure (T3). Hemolysis will be assessed in all three samples 1) using flow cytometry (by means of measurement of "erythrocyte microparticles detected by the presence of antigens glycophorin A and Annexin V) and 2) using ELISA method (assessment of "cell free hemoglobin " concentration). Additionelly, standard biochemistry and blood count analysis will be done from the T1 and T3 samples (the concentration of lactate dehydrogenase, haptoglobin, indirect bilirubin, reticulocytes, and immature reticulocyte fraction).

Primary hypothesis is that the level of hemolysis will be higher after PF ablation compared to RF ablation. Since no studies were published on the hemolysis either during RF or PF ablation, no reliable power calculation can be done.

ELIGIBILITY:
Inclusion Criteria:

* symptomatic atrial fibrillation indicated for catheter ablation
* willingness to participate

Exclusion Criteria:

* pregnancy
* any known malignant or non-malignant hematological disorder
* malignancy
* age > 75 years
* any disease associated with hemolysis
* hemoglobin concentration less than 100 g/L
* liver cirrhosis

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with symptomatic paroxysmal or non-paroxysmal atrial fibrillation indicated according current guideliens for the cathter ablation of atrial fibrillation, i.e. pulmonary vein isolation
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2023-11-15 (Estimated); Primary Completion 2024-03-30 (Estimated); Study Completion 2024-03-30 (Estimated)

PRIMARY OUTCOMES:
Erythrocyte (red blood cells, RBC) microparticles | One day after the procedure
  The concentration of erythrocyte microparticles /µL. Analysis using flow cytometry, as the concentration of total erythrocyte mictoparticles in platelet-rich plasma.
Cell free hemoglobin | One day after the procedure
  The concentration of cell-free hemoglobin, using ELISA measurement, in g/L

SECONDARY OUTCOMES:
Lactate-dehydrogenase | One day after the procedure
  The concentration of lactate-dehydrogenase (µkat/L)
Haptoglobin | One day after the procedure
  The concentration of haptoglobin (g/L)
Indirect bilirubin | One day after the procedure
  The concentration of indirect bilirubin (µmol/L)
Reticulocytes | One day after the procedure
  The absolute concentration of reticulocytes
Immature reticulocyte fraction (IRF) | One day after the procedure
  The percentage of immature reticulocytes of all reticulocytes (%)

CONTACTS AND LOCATIONS:
Locations (1):
- Cardiocenter, 3rd Medical School, Charles University and University Hospital Kralovske Vinohrady, Prague, Czechia

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared based on individual request
Supporting Information: CSR
Time Frame: Starting after the publication of results
Access Criteria: By request on PI

REFERENCES:
- [Result] Zoni-Berisso M, Filippi A, Landolina M, Brignoli O, D'Ambrosio G, Maglia G, Grimaldi M, Ermini G. Frequency, patient characteristics, treatment strategies, and resource usage of atrial fibrillation (from the Italian Survey of Atrial Fibrillation Management [ISAF] study). Am J Cardiol. 2013 Mar 1;111(5):705-11. doi: 10.1016/j.amjcard.2012.11.026. Epub 2012 Dec 28. PMID 23273528
- [Result] Reddy VY, Dukkipati SR, Neuzil P, Anic A, Petru J, Funasako M, Cochet H, Minami K, Breskovic T, Sikiric I, Sediva L, Chovanec M, Koruth J, Jais P. Pulsed Field Ablation of Paroxysmal Atrial Fibrillation: 1-Year Outcomes of IMPULSE, PEFCAT, and PEFCAT II. JACC Clin Electrophysiol. 2021 May;7(5):614-627. doi: 10.1016/j.jacep.2021.02.014. Epub 2021 Apr 28. PMID 33933412
- [Result] Ekanem E, Reddy VY, Schmidt B, Reichlin T, Neven K, Metzner A, Hansen J, Blaauw Y, Maury P, Arentz T, Sommer P, Anic A, Anselme F, Boveda S, Deneke T, Willems S, van der Voort P, Tilz R, Funasako M, Scherr D, Wakili R, Steven D, Kautzner J, Vijgen J, Jais P, Petru J, Chun J, Roten L, Futing A, Rillig A, Mulder BA, Johannessen A, Rollin A, Lehrmann H, Sohns C, Jurisic Z, Savoure A, Combes S, Nentwich K, Gunawardene M, Ouss A, Kirstein B, Manninger M, Bohnen JE, Sultan A, Peichl P, Koopman P, Derval N, Turagam MK, Neuzil P; MANIFEST-PF Cooperative. Multi-national survey on the methods, efficacy, and safety on the post-approval clinical use of pulsed field ablation (MANIFEST-PF). Europace. 2022 Sep 1;24(8):1256-1266. doi: 10.1093/europace/euac050. PMID 35647644
- [Result] Liu D, Li Y, Zhao Q. Effects of Inflammatory Cell Death Caused by Catheter Ablation on Atrial Fibrillation. J Inflamm Res. 2023 Aug 17;16:3491-3508. doi: 10.2147/JIR.S422002. eCollection 2023. PMID 37608882